CLINICAL TRIAL: NCT02533531
Title: Proof of Concept Study for 1 Lead Patch Technology
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was halted to make device updates
Sponsor: LifeWatch Services, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CIP-F010
Record Dates: First submitted 2015-08-25; First posted 2015-08-26 (Estimated); Results first posted 2018-04-06 (Actual); Last update posted 2018-04-06 (Actual); Status verified 2018-03

CONDITIONS: Telemetry

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- 1-Lead Outpatient Telemetry (Experimental): 1-Lead Outpatient Patch study participants. Patients assigned to outpatient telemetry monitoring will receive the 1-Lead patch upon discharge from hospital inpatient status. ECG data will be submitted by the 1-lead patch to a central database.
  Interventions: Device: 1-Lead Patch

INTERVENTIONS:
Device: 1-Lead Patch — The 1-Lead Patch will record and transmit ECG data to a gateway, which will then transmit the data to a central database.

SUMMARY:
This study is intended to assess the feasibility and usability of the 1 Lead Patch as a whole, on patients outside the hospital, in the out-patient setting.

DETAILED DESCRIPTION:
This study is a two-phase evaluation of the use of a 1 Lead Patch System to monitor electrocardiogram (ECG) data and send the data to the LifeWatch Service Center, in the same manner as the existing ACT ambulatory telemetry system. It will be used in parallel with the standard 3 Lead ACT testing equipment used to monitor ECG outside the hospital. This study will not address safety or effectiveness and no comparator groups will be used. This study will not be treating any particular disease or condition and no randomization or blinding is required. Subjects will be selected in conjunction with their need for current outpatient telemetry monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female referred for 3 Lead ACT monitoring for between 7 and 14 days.
* Be recently prescribed a LifeWatch 3 Lead ACT monitor

Exclusion Criteria:

* under 21-years old
* pregnant or who may become become pregnant during the investigation period
* using internal or external defibrillators
* who are using pacemakers or implantable loop recorders
* showing skin damage on the chest, such as burns, irritation, infections, wounds, etc.
* meeting any contraindications for a patch biosensor

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2014-04-16 (Actual); Primary Completion 2016-06-09 (Actual); Study Completion 2016-06-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vivek Reddy, MD FACC FHRS, Principal Investigator — Mt. Sinai Medical Center; Marie Noelle-Langan, MD, Principal Investigator — Mt. Sinai Medical Center
Locations (1):
- Mt. Sinai Medical Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 1-Lead Outpatient Telemetry
Started | 1
Completed | 0
Not Completed | 1
Not completed — Device did not turn on | 1

BASELINE CHARACTERISTICS:
Population: The single enrolled subject did not complete study procedure. Therefore no analysis was completed.
Arm/Group | 1-Lead Outpatient Telemetry
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants] — Population: The single enrolled subject did not complete study procedure. Therefore no data was collected / analyzed.
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The single enrolled subject did not complete study procedure. Therefore no data was collected / analyzed.
Region of Enrollment [Number; unit: participants] — Population: The single enrolled subject did not complete study procedure. Therefore no data was collected / analyzed.

OUTCOME MEASURES:

1. Primary Outcome: Composite Outcome Measure - 100% Successful ECG Acquisition
Description: Successful acquisition of ECG data by the 1-Lead patch with transmission to the central database via the gateway. Each patch includes a 'brain' that collects the ECG data and then transmits it to a cellular device called the 'gateway'. The gateway uses the cellular network to transmit the data to the central database. This is a composite outcome measure. Data were not collected.
Time Frame: Between 7 and 14 days
Population: Data were not collected.
Arm/Group | 1-Lead Outpatient Telemetry
Number analyzed (Participants) | 0

2. Secondary Outcome: Composite Outcome Measure - Adhesive Performance - Measurement of Skin Irritation Resulting From Adhesive Used With 1-Lead Patch
Description: Successful performance of the 1-Lead Patch adhesive throughout the study period for each subject. Subject skin irritation will be assessed upon initial placement of the 1-Lead Patch by the clinical caregiver. Subjects will be asked to self-assess skin irritation and to report to the clinician at the end of the trail period. Data were not collected.
Time Frame: Between 7 and 14 days
Population: Data were not collected.
Arm/Group | 1-Lead Outpatient Telemetry
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | 1-Lead Outpatient Telemetry
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No